CLINICAL TRIAL: NCT06489899
Title: Peer Education for Gender Inclusion and Substance Use in Southern Africa (PEGISUS): A Pilot Trial Testing a Peer-based Intervention in Vocational Training Programs
Brief Title: Peer Education for Gender Inclusion and Substance Use in Southern Africa
Acronym: PEGISUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: SolidarMed (Other); University of Zambia (Other); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AO202300095
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Substance Use; Gender Role
Keywords: gender; substance use; Zimbabwe; Zambia; South Africa
MeSH Terms: conditions — Substance-Related Disorders; Coitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEGISUS (Experimental): PEGISUS is based on two existing evidence-based interventions: Reducing Alcohol and Drug use and other Problem behavior in Adolescent Learners (RAD-PAL) and Manhood 2.0. RAD-PAL was developed to target primary substance use and other challenging behaviors. Manhood 2.0 was developed to reduce traditional gender beliefs. These interventions have been adapted based on formative work with the target user group. PEGISUS will be embedded into existing vocational training programs and delivered by existing staff at these institutions.
  Interventions: Behavioral: PEGISUS
- Standard of Care (No Intervention): Standard of care is receiving the vocational training program that is offered through the partner organization and a healthcare referral for substance use. The vocational training programs are SOZO Foundation (South Africa), Build It International (Zambia), and Masvingo Polytechnic (Zimbabwe). SOZO Foundation offers training in six different vocational areas, including hairstyling, coding, and nutrition. They also teach life skills. Build It International offers construction programs and support beyond initial training through connection to employment and mentorship. Masvingo Polytechnic offers many programs, including electrical engineering, welding, guidance counseling, motor mechanics, and catering.

INTERVENTIONS:
Behavioral: PEGISUS — PEGISUS is an 8-session intervention for substance use and gender equitable beliefs.
  Other Names: Peer Education for Gender Inclusion and Substance Use in Southern Africa
  Arms: PEGISUS

SUMMARY:
The goal of this trial is to test the effectiveness of a brief, behavioral peer group intervention called "PEGISUS" (Peer Education for Gender Inclusion and Substance Use in Southern Africa), on substance use, which will be embedded within existing vocational training programs in Zambia, Zimbabwe, and South Africa. Established peer groups who receive the PEGISUS intervention will complete nine sessions of an adapted intervention for substance use and gender equitable beliefs, embedded into vocational training programs. This will be compared to a standard of care control condition, which involves the vocational training program that is offered through the partner organization and a healthcare referral for substance use. The vocational training program partners are Sozo Foundation (South Africa), BuildIt International (Zambia), and Masvingo Polytechnic (Zimbabwe). Participants in both conditions will complete assessments at baseline, 12-weeks follow-up, and 24-weeks follow-up, consisting of self-reported questionnaires.

DETAILED DESCRIPTION:
Adolescents and young adults (AYA) make up a large proportion of the population in sub-Saharan Africa (SSA), including in South Africa, Zambia, and Zimbabwe, but also face increasingly high levels of disability and mortality. This is influenced by high levels of substance use and occurs in a predominantly gender normative environment that places young men, women, and non-cisgender young people at risk. One of the primary risk factors for AYA substance use is having peers who also engage in substance use, however, treatments do not target peers. Adoption of traditional gender norms that favor men are also associated with worse health outcomes for both genders. For AYA boys/men, this includes substance use, sexual risk-taking behaviours, and engaging in intimate partner violence; for AYA girls/women, there is increased risk of acquiring sexually transmitted infections and HIV as well as poor educational attainment, such as school dropout. It is necessary to target such gender norms to improve health outcomes of both genders. Addressing these traditional gender beliefs during the AYA period may be more impactful than during adulthood. AYA education and/or vocational training (VT) programs increase chances for a successful future in a setting where employment of youth is generally low. Overall, key behaviors during the AYA period in SSA support well-being across the lifespan, including educational/ vocational attainment, developing healthy coping beyond substance use, and adoption of equitable gender norms. This study seeks to test a brief, behavioral intervention focused on substance use reduction and development of equitable gender norms, which will be delivered to peer groups enrolled in existing VT programs in South Africa, Zambia, and Zimbabwe.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults 16 - 24 years old
* At least weekly self-reported alcohol/drug use in a peer group in the past month or at least monthly heavy episodic drinking with peers over the past three months
* Comfortable communicating in the predominant local language or English
* Lives in the target community and plans to remain in the area for the next 12 months
* Eligible to participate in the vocational training (VT) program (according to the VT program's own entry guidelines) and willing to participate in the entirety of the program
* Interested to participate in a substance reduction and gender equity beliefs program and able to identify 2 to 5 peers to join
* Willing to have PEGISUS workshop sessions audio/video-recorded (if assigned to that group)

Exclusion Criteria:

* Untreated major mental illness that interferes with study participation, such as active suicidality, or unmanaged bipolar disorder or psychotic disorder
* Currently receiving psychological treatment for substance use
* Participation in another VT/skills development program or another trial that is judged by the site investigator as non-compatible with this study
* Unable to provide informed consent or informed assent

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Self-reported substance use for participants aged 18 and older | Change from baseline to 12-week follow-up assessment [range ≥8-20 weeks]
  Self-report using the Alcohol, Smoking and Substance involvement Screening Test (ASSIST; for participants aged 18 and older). Higher scores indicate more substance use and associated problems.
Self-reported substance use for participants aged 16 and 17 | Change from baseline to 12-week follow-up assessment [range ≥8-20 weeks]
  Self-report using the Alcohol, Smoking and Substance Involvement Screening Test for Youth (ASSIST-Y; for participants aged 16 and 17). Higher scores indicate more substance use and associated problems.

SECONDARY OUTCOMES:
Self-reported substance use for participants aged 18 and older | Change from baseline to 24-week follow-up assessment [range >20-32 weeks]
  Self-report using the Alcohol, Smoking and Substance involvement Screening Test (ASSIST; for participants aged 18 and older). Higher scores indicate more substance use and associated problems.
Self-reported substance use for participants aged 16 and 17 | Change from baseline to 24-week follow-up assessment [range >20-32 weeks]
  Self-report using the Alcohol, Smoking and Substance Involvement Screening Test for Youth (ASSIST-Y; for participants aged 16 and 17). Higher scores indicate more substance use and associated problems.
Self-reported gender equitable beliefs | Change from baseline to 12-week follow-up assessment [range ≥8-20 weeks] and 24-week follow-up assessment [range >20-32 weeks]
  Self-report using the adapted 23-item version of the Gender Equitable Men's Scale. Items are scored on a 3-point likert scale with higher scores representing more equitable norms.
Attendance at vocational training program | 24-week follow-up assessment [range >20-32 weeks]
  Number of months of attendance in vocational training program.
Rate of completion of vocational program | 24-week follow-up assessment [range >20-32 weeks]
  Number and percentage of participants that completed the vocational training program.
Employment | 24-week follow-up assessment [range >20-32 weeks]
  Subsequent employment status will be taken from vocational training program records, supplemented with self-report.
Income earned | 24-week follow-up assessment [range >20-32 weeks]
  Income earned will be taken from vocational training program records, supplemented with self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Belus, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (3):
- SOZO Foundation, Cape Town, Western Cape, South Africa
- Build It International, Chibombo, Zambia
- Masvingo Polytechnic, Masvingo, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized data and statistical code will be deposited alongside the published peer-reviewed papers, in alignment with data sharing and verification procedures. Other investigators wishing to access the data for additional analyses can contact the study PI so that the appropriate documents (e.g., data sharing, ethics approvals) can be arranged.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: A de-identified dataset will be deposited in an open-access data repository at the end of the project and once the objectives specified in the protocol have been addressed.
Access Criteria: The data can be accessed by the public, through creation of an account with Open Science Foundation, an open-access data repository.

REFERENCES:
- [Background] Carney T, Johnson K, Carrico A, Myers B. Acceptability and feasibility of a brief substance use intervention for adolescents in Cape Town, South Africa: A pilot study. Int J Psychol. 2020 Dec;55(6):1016-1025. doi: 10.1002/ijop.12668. Epub 2020 Apr 13. PMID 32285449
- See also: Program overview and final results of Manhood 2.0's effects on gender equitable beliefs — https://www.equimundo.org/wp-content/uploads/2019/06/PM-Manhood-2-0-Program-Overview-v1-7-E.pdf